CLINICAL TRIAL: NCT02245243
Title: An Open Label Evaluation of the Single Dose Pharmacokinetics of Delafloxacin in Subjects With and Without Hepatic Impairment
Brief Title: Pharmacokinetics of Delafloxacin in Subjects With and Without Hepatic Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Melinta Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML-3341-112
Record Dates: First submitted 2014-09-17; First posted 2014-09-19 (Estimated); Last update posted 2015-04-30 (Estimated); Status verified 2015-04

CONDITIONS: Hepatic Impairment
Keywords: Hepatic Impairment, single dose, intravenous
MeSH Terms: interventions — delafloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Delafloxacin (Experimental): Single Dose 300 mg IV
  Interventions: Drug: Delafloxacin

INTERVENTIONS:
Drug: Delafloxacin — Plasma pharmacokinetic parameters: AUC0-t, AUC0 inf, Cmax, Tmax, λz, t1/2, MRTinf, CL, CLnr, Vss, Vz

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetic profile, safety, and tolerability of a single intravenous (IV) dose of delafloxacin in normal healthy subjects and subjects with mild, moderate, or severe hepatic impairment.

DETAILED DESCRIPTION:
pharmacokinetic profile, safety, and tolerability of a single intravenous (IV) dose of delafloxacin in normal healthy subjects and subjects with mild, moderate, or severe hepatic impairment. AUC0-t, AUC0 inf, Cmax, Tmax, λz, t1/2, MRTinf, CL, CLnr, Vss, Vz

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) between 18.5 and 40 kg/m2, inclusive.
* Able to provide written, informed consent before initiation of any study related procedures, and is able, in the opinion of the investigator, to comply with all the requirements of the study.

Hepatically Impaired Subjects Only (Groups A, B, and C):

-Has a clinical diagnosis of cirrhosis and has been classified as having mild (Group A), moderate (Group B), or severe (Group C) hepatic impairment as defined by the Child-Pugh classification system (Section 7.2).

Healthy Subjects Only (Group D):

-Must be in good health as determined by the investigator based on medical history, clinical laboratory results, vital sign measurements, 12 lead electrocardiogram [ECG] results, and physical examination findings

Exclusion Criteria:

* All Subjects (Groups A through D):
* Has a clinically significant abnormality in past medical history or at the screening physical examination (excluding hepatic impairment and other related stable medical conditions within the hepatically impaired population of subjects) that in the investigator's or sponsor's opinion may place the subject at risk or interfere with outcome variables of the study. This includes, but is not limited to, history or current cardiac, renal, neurologic, gastrointestinal, respiratory, hematologic, or immunologic disease.
* History or presence of an abnormal ECG that, in the investigator's opinion, is clinically significant and would preclude study participation.
* Has any surgical or medical condition (active or chronic) that may interfere with drug absorption, distribution, metabolism, or excretion of the study drug, or any other condition that may place the subject at risk (history of cholecystectomy is allowed).
* Has a functioning liver transplant
* Has a history of drug and/or alcohol abuse within 6 months before Screening
* Has a history of or current clinically significant mental disorder or an antagonistic personality that compromises the validity of the informed consent.
* Has donated blood or plasma within 30 days before dosing, or has lost more than 1200 mL of blood within 4 months before the first dose of study drug.
* Has a history of AIDS or subject has positive results for HIV at Screening.

Hepatically Impaired Subjects Only (Groups A, B, and C):

* Has had clinical exacerbation of liver disease within 14 days before study drug administration (eg, abdominal pain, ascites, nausea, vomiting, anorexia, fever, or worsening of laboratory results related to hepatic function).
* Has evidence of acute viral hepatitis within 1 month before Day -1, has clinically demonstrable massive tense ascites, has evidence of severe or acute renal failure, has active stage 3 or stage 4 encephalopathy.

Healthy Subjects Only (Group D):

-Has a positive test result for hepatitis B surface antigen or hepatitis C virus antibody.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-09; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Plasma pharmacokinetic parameters: • AUC0-t, AUC0 inf, Cmax, Tmax, λz, t1/2, MRTinf, CL, CLnr, Vss, Vz | Baseline through 72 hours post-dose

SECONDARY OUTCOMES:
Safety endpoints: AEs, clinical laboratory results (serum chemistry, coagulation, hematology, and urinalysis), vital sign measurements, 12-lead ECG measurements, and physical examination findings | Baseline through 72 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Sue K Cammarata, MD, Study Director — CMO, MelintaTtherapeutics, Inc.
Locations (2):
- United States (2):
  - Melinta 112 Study Site, Miami, Florida
  - Melinta 112 Study Site, Orlando, Florida

REFERENCES:
- [Derived] Hoover R, Marbury TC, Preston RA, Quintas M, Lawrence LE, Paulson SK, Luke DR, Cammarata SK. Clinical Pharmacology of Delafloxacin in Patients With Hepatic Impairment. J Clin Pharmacol. 2017 Mar;57(3):328-335. doi: 10.1002/jcph.817. Epub 2016 Oct 14. PMID 27570245